CLINICAL TRIAL: NCT02982551
Title: Insulin Modulation of fMRI Connectivity and Food Reward
Brief Title: Insulin Modulation of fMRI Connectivity in Healthy Adults
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Principal Investigator Departed University
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John Patrick Ryan, PhD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO15040502
Record Dates: First submitted 2016-11-22; First posted 2016-12-05 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Insulin; Magnetic Resonance Spectroscopy; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperinsulinemic Clamp (Experimental): Participants will complete two MRI scans approximately one hour apart - one under baseline conditions and the second during an insulin infusion. Each scan will include data collected during rest, and a taste task. The taste task involves receiving milkshake or a tasteless solution. After the first scan, an isoglycemic-hyperinsulinemic clamp will be implemented. An IV will be placed in the antecubital vein of of arm for infusion of insulin and dextrose. HumuLIN®-R regular insulin will be infused at 40 mU/m2/min. A second IV will be inserted in the back of the hand on the opposite arm to allow for frequent sampling of blood glucose levels. Dextrose infusion will be used to keep the blood sugar level within 5mg/dl of the baseline value. The study team will monitor blood glucose levels and adjust dextrose infusions as necessary. Thirty minutes after starting the insulin infusion, participants will be moved back into the bore of the MRI scanner for the repeat scans.
  Interventions: Drug: Insulin; Other: Taste Task; Other: Magnetic Resonance Imaging; Drug: Dextrose

INTERVENTIONS:
Drug: Insulin — Insulin will be administered peripherally to observe the effects of circulating insulin on brain activity
  Other Names: HumuLIN®-R
Other: Taste Task — Participants will taste milkshakes and a tasteless solution to observe the brain responses to palatable taste.
Other: Magnetic Resonance Imaging — Participants will complete two MRI scans approximately 60 minutes apart - one under baseline fasting conditions and the second during isoglycemic-hyperinsulinemia. Each functional scan will include a resting-state BOLD sequence followed by a taste-reward task. Functional MRI sequences will last approximately 30 minutes. MRI scanning will also include approximately 30 minutes of structural MRI scans.
Drug: Dextrose — During hyperinsulinemic clamp, participants will be infused with a variable rate dextrose infusion will be used to keep the blood sugar level within 5mg/dl of the baseline glucose value.

SUMMARY:
This study evaluates the effects of changing insulin levels on brain activity. Participants will complete functional magnetic resonance imaging (fMRI) scans during fasting conditions, then during an insulin infusion.

DETAILED DESCRIPTION:
Insulin is a hormone released by the pancreas in response to increases in glucose levels that result from food intake. In addition to stimulating glucose uptake in the periphery, insulin signals the central nervous system to induce satiety and inhibit feeding behavior.

To begin to identify the specific effects of circulating insulin on brain networks, the current study will recruit healthy participants who will undergo two functional magnetic resonance imaging scans. One scan will be performed in the fasted state, and the alternate scan will be conducted during an isoglycemic hyperinsulinemic clamp.

This project will allow us to identify the specific effects of circulating insulin on brain reactivity to palatable food.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 24
* HOMA-IR < 1.55 (homeostatic model assessment of insulin resistance - ((glucose x insulin) / 405)).

Exclusion Criteria:

* Current or lifetime history of any cardiovascular disease or surgery (including hypertension, stroke, myocardial infarction, congestive heart failure, atrial or ventricular arrhythmias, coronary bypass, carotid artery, or peripheral vascular surgery)
* Current or lifetime history of cancer, a chronic kidney or liver condition, type I or II diabetes, or any pulmonary or respiratory disease
* Current or lifetime diagnoses of any substance abuse
* Positive urine drug screen
* Current or lifetime use of glucocorticoid medications for >1 month
* A previous cerebrovascular accident or trauma involving loss of consciousness
* Previous neurosurgery or history of a neurological condition
* Pregnancy (females)
* Claustrophobia
* Ferrous metallic implants or any surgically placed medical device not cleared for safety at 3Tesla MRI strength
* Peripheral vascular disease
* Liver, kidney, or active blood disease
* Peripheral neuropathy
* Anemia (hematocrit <34%)
* Inability and/or willingness to comply with the protocol as written
* Fasting glucose > 126 mg/dL
* Currently taking blood thinners such as coumadin, Lovenox, etc.
* Currently taking any medications that can alter glucose homeostasis (steroids, glucocorticoids, nicotinic acid)
* Current use of any psychotropic medications (SSRI, SNRI, etc.)
* Currently taking thiazolidinediones or insulin
* Currently use of statins or anti-hypertensive medications
* Use of medications related to HIV that can affect insulin sensitivity. We will NOT specifically test for HIV serostatus.
* Females currently on hormone replacement therapy (HRT) less than 6 months
* Participants will be instructed to abstain from eating, drinking (other than water), smoking and exercise for the 12 hours prior to each study visit.
* Being left handed
* Body mass index above 24 or below 18
* Milk allergy / lactose intolerance
* Polycystic ovary syndrome

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
fMRI BOLD Response in Brain | During Taste Task in fMRI Scanner. Task Duration is approximately 14 minutes.
  The investigators will monitor the blood oxygen level dependent response using fMRI and compare activation during "taste" trials vs. "no taste" trials.

CONTACTS AND LOCATIONS:
Overall Officials: John P Ryan, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No